CLINICAL TRIAL: NCT02630173
Title: Evaluation of Endodontic Status on Periodontal Healing of Concomitant Endodontic Periodontal Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, Proffesor and Head, Postgraduate Institute of Dental Sciences Rohtak
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PGIDS/IEC/2014/111
Record Dates: First submitted 2015-12-06; First posted 2015-12-15 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Periodontal Pocket
Keywords: endodontic treatment; scaling; root planning
MeSH Terms: conditions — Periodontal Pocket | interventions — Tooth Exfoliation; Root Planing; Endodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non vital teeth with apical radiolucency (Experimental): Endodontic treatment was performed in non vital teeth with periapical radiolucency. Local anesthesia was provided (2% Novocaine with 1:80,000 epinephrine), isolation with rubber dam and standard access cavity preparation was done.Using 3 % sodium hypochlorite, canal negotiation was done & apical patency was achieved with #10 or #15K-files. Coronal flaring with # 2 and #3 Gates-Glidden drills was done.Calcium hydroxide was filled in the canals with the help of a lentulo spiral.At the second appointment,calcium hydroxide paste was removed and copious irrigation with 3% sodium hypochlorite was followed by 5.0 mL 17% ethylenediaminetetraacetic acid with a final rinse of 5.0 mL of 3% sodium hypochlorite. The canals were obturated with gutta-percha and ZOE sealer.
  Interventions: Procedure: Scaling and root planing; Other: Endodontic treatment
- Vital teeth (Active Comparator): Only scaling and root planing will be done in contralateral vital tooth with pocket depth >5mm .Non surgical periodontal treatment in the form of scaling and root planing was provided in minimum of two sessions using ultrasonic scaler (Satelec P5 Booster Suprasson) and hand instruments (Hu-friedy scalers and curettes).
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — Scaling and root planing was done in both the groups
  Other Names: Non surgical Periodontal treatment
Other: Endodontic treatment — In non vital teethRoot canal treatment was completed in two visits. 3% Naocle was used as irritant and calcium hydroxide was used as intracanal medicament .Obturation was done with gutta percha.
  Other Names: root canal treatment
  Arms: Non vital teeth with apical radiolucency

SUMMARY:
Introduction:

To evaluate the effect of untreated endodontic infection on periodontal status in untreated non vital teeth with periapical radiolucency as compared to contralateral vital teeth. And also to evaluate the role of endodontic treatment on periodontal healing in successfully endodontically treated teeth with contralateral vital teeth.

Methods:

This study was performed in two parts. First part of this study was an observational cross sectional survey and second part was a clinical trial on patients selected from the survey.

DETAILED DESCRIPTION:
Title: EVALUATION OF ENDODONTIC STATUS ON PERIODONTAL HEALING OF CONCOMITANT ENDODONTIC PERIODONTAL LESIONS

INTRODUCTION:

Although deleterious effects of endodontic tissue on the periodontium are well documented, the converse effect of periodontal disease on pulp remains unclear. There is abundance of research on the avenues of communication but still many doubts exist. High prevalence of accessory canals has been seen but not all primary endodontic lesions drain through the periodontal ligament. Many endodontic lesions are more prone to drain through cortical bone rather than through the periodontal ligament. It may be because of the nature of periradicular lesions which initially try to expand horizontally through cancellous bone and then progressing vertically. Evidence also suggests that endodontically treated teeth lack the same proprioceptive capability as endodontically untreated teeth so they may be subjected to greater occlusal forces. More forces could enhance the propagation of fracture lines along the root surface, resulting in more periodontal attachment loss. Also teeth associated with either root perforations or fractures appear to follow periodontal drainage routes whereas lesions of primarily pulpal origin seem to remain localized or drain through cortical bone. Many explanations are provided, firstly periodontal ligament may be resistant to bacterial insult of endodontic origin, or injuries originating through mechanical trauma are faintly recognized, causing a subtle attachment loss occurring secondary to routine endodontic disease. Another explanation could be that the main or accessory canals might not be the solo and most important route of communication and endodontic infection might also proceed along cervically located dentinal tubules.

A group of retrospective and experimental studies in the past demonstrated the effect of endodontic infection on periodontal status and healing. A series of retrospective studies performed on single rooted teeth of periodontitis prone patients correlated endodontic infection with periodontal status in terms of pocket depth and attachment loss. Teeth with periapical radiolucency demonstrated deeper pockets and more radio graphic attachment loss as compared to a healthy tooth. Non surgical periodontal treatment with horizontal defects depicted reduced mean pocket depth reduction and increased radio graphic attachment loss in teeth with periapical pathology in comparison with endodontically intact tooth. Even multi rooted teeth with periapical destruction in periodontitis prone patients exhibited significantly greater mean probing depth compared to teeth without periapical destruction. Mandibular molars with periapical destruction showed ≥ 3 mm horizontal furcation depth. In all these studies periodontal parameters of teeth (either root filled or with a periapical radiolucency) were compared with an endodontically intact tooth also present in the patients without any consideration of quality of obturation.

Research has denoted that endodontic treatment influences the periodontal healing and periodontal status of tooth.

Reduced healing potential of the periodontal structures by endodontic treatment was evident in human studies.

Endodontic infection is a local modifying risk factor is based on retrospective studies experimental studies. Prospective studies have been carried out to evaluate effect of endodontic treatment on periodontal healing only. The present understanding on the effect of endodontic status on periodontal status and healing is mainly based on retrospective studies where numbers of variables evaluated are limited with a low level of reliability. They lack the power to accept or reject any hypothesis. The retrospective studies had no control on quality of obturation and lacked standardization of radiographs. Moreover the experimental studies were conducted in extreme conditions and lacked similarity to clinical conditions. No prospective study has yet compared the periodontal status as well as periodontal healing in untreated non vital teeth and successfully endodontically treated teeth with contralateral vital teeth.

So, the purpose of this study was to evaluate the effect of untreated endodontic infection on periodontal status in untreated non vital teeth with periapical radiolucency as compared to contralateral vital teeth. And also to evaluate the role of endodontic treatment on periodontal healing in successfully endodontically treated teeth with contralateral vital teeth.

Methods:

All patients with the diagnosis of generalized chronic periodontitis were screened for a non vital tooth with periapical radiolucency that also had contralateral vital tooth with normal periapical conditions in the radio graph. A split mouth design was followed with non vital tooth with periapical radiolucency (test group 1) and a contralateral vital tooth (test group2) present in each patient.

Parameters recorded:

1. Site specific clinical parameters like probing depth, clinical attachment loss, bleeding on probing, plaque score.
2. Digital radio graphic evaluation was done by taking intra oral periapical radiographs. Bone level and periapical score was recorded.

Follow up of patients was done at 1, 3 and 6 months to evaluate the improvement in periodontal parameters and PAI score.

Endodontic treatment protocol: Using a standardized protocol root canal treatment was performed by a single operator for all cases. Initially local anesthesia was provided (2% Novocaine with 1:80,000 epinephrine), isolation was achieved by rubber dam and standard access cavity preparation was done.

Using 3 % sodium hypochlorite, canal negotiation was done & apical patency was achieved with #10 or #15K-files. Coronal flaring was created with # 2 and #3 Gates-Glidden drills (Dentsply Maillefer, Tulsa, OK). With the help of a Root-ZX apex locator working length of each canal was established (J Morita, Irwine, CA) and then verified with radiographs.

A crown down technique for canal instrumentation was followed using hand K files. The master apical file size was set at 3 sizes larger than the first binding file at working length. Instrumentation was accompanied with copious irrigation of 3% sodium hypochlorite using 27 gauge needles. Calcium hydroxide was filled in the canals with the help of a lentulo spiral and patients were scheduled for a second appointment to complete root canal therapy within 10 days to obturate the canal. At the second appointment, after removing the calcium hydroxide paste circumferential filing with Hedstrom-type files was done and copious irrigation with 3% sodium hypochlorite was followed by 5.0 ml 17% ethylenediaminetetraacetic acid with a final rinse of 5.0 ml of 3% sodium hypochlorite.

The canals were dried with sterile paper points and obturated by using lateral condensation technique with gutta-percha (Dentsply Tulsa Dental) and ZOE sealer.

Periodontal treatment protocol - Non surgical periodontal treatment in the form of scaling and root planing was provided in minimum of two sessions using ultrasonic scaler (Satelec P5 Booster Suprasson) and hand instruments (Hu-friedy scalers and curettes). In the first session supragingival scaling was done and in the second session root planing was performed until a clinically hard, smooth surface was achieved.

Sample size:

Assuming the effect size of 0.5, power .95 and α=0.05 a sample of 105 patients in each group was required for the survey to show clinically significant difference. For the clinical trial with the effect size of 1, power .80 and α=0.05, 17 patients in each group were required to elicit a clinical significant difference. To further compensate for the drop outs, 28 patients in each group were enrolled for the study.

Statistical Analyses:

Shapiro-Wilk normality test showed that data for the survey and for the clinical trial was non normally distributed. The differences between the groups in survey and the clinical trial for continuous variables were assessed using Mann-Whitney U test and for categorical variables (brushing habits and dexterity) using chi square (χ2) test.

Partial correlation between variables in the survey was assessed after controlling the potential confounders like age and PI. Multiple linear regression analysis was used to develop models of predictor variables (PAI, tooth, gender) associating to the dependent variables (mean probing depth (PD), maximum probing depth (PD max), mean attachment loss (AL), maximum attachment loss (AL max), mean bone level. Scoring of pocket depth, attachment loss and PAI was further categorized as 0 (PD<4mm, AL<4mm and PAI=absence of radiolucency) and 1 (≥4 to ≤8 PD, AL and PAI=presence of radiolucency). Similarly scoring of mean bone level was categorized as 0 (<5mm) and 1 (≥5mm) for purpose of logistic regression. The evaluation of the association between PD, AL and PAI was estimated by odds ratio (OR) and 95% confidence intervals (95% CI).

Evaluation of improvement in clinical parameters (PD, PD max, AL, AL max, BOP, PI, PAI) in the two test groups (Test group1 and Test group 2) was done using intra group comparison at baseline to 1month, baseline to 3 months, baseline to 6 months,1 to 3 months, and 3-6 months using the Wilcoxon signed rank test. The differences in improvement of clinical parameters between the two test groups ((Test group1 and Test group 2) was assessed using Mann-Whitney-U analysis. Statistical signiﬁcance was set at the 95% probability level (P < .05).

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than or equal to18 years with more than 20 remaining teeth.
2. Generalized chronic periodontitis was considered when ≥30% of sites were involved with clinical attachment loss (CAL) slight =1 or 2 mm, Moderate =3 or 4 mm, and Severe ≥5 mm41.
3. Non vital tooth and contralateral vital tooth with PD ≥ 5 mm on at least one site.
4. Non vital tooth confirmed by electric pulp test and cold test.
5. Contralateral tooth with normal periapical conditions in the radiograph and with no evidence of root canal treatment and was vital as confirmed by electric pulp test and cold test.

Exclusion Criteria:

1. Patients younger than 18 years
2. Non vital tooth and contralateral vital tooth with mean PD>8 and<4.
3. Endodontically treated teeth
4. Smokers
5. Unrestorable teeth
6. Contralateral tooth having proximal carious lesions or was non vital.
7. Inflammatory root resorption
8. Fractured / Perforated roots
9. Serious medical illness; Patients with uncontrolled or poorly controlled diabetes, unstable or life threatening conditions or requiring antibiotic prophylaxis (including infective endocarditis or prosthetic joint prophylaxis and immune compromising disorder)
10. Pregnant mothers
11. A history of recent periodontal therapy (with in previous 6 months)
12. Teeth with established endodontic-periodontal lesion exhibiting less than 2 mm radiopaque bone between the periapical lesion and periodontal destruction, in which the periodontal probe reached the apex.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Improvement in periodontal parameters Probing depth | baseline to 6months
  periodontal parameters pocket depth (in mm) was measured at baseline to 6 months with the help of calibrated manual periodontal probe.

SECONDARY OUTCOMES:
plaque score | baseline to 6 months
bleeding on probing | baseline to 6 months
periapical score | baseline to 6 months
attachment loss | baseline to 6 months
  using a calibrated manual periodontal probe in mm.